CLINICAL TRIAL: NCT03660306
Title: Observational Study Evaluating the Impact of Opioid Free Anesthesia During Lung Protective Ventilation on Postoperative Oxygen Saturation.
Brief Title: Impact of OFA During LPV on Postoperative Oxygen Saturation
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, MD PhD, AZ Sint-Jan AV
Other Study IDs: OS impact OFA on SAT d LPV
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Decreased Lung Compliance; Oxygen Requirement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- opioid anesthesia: classical anesthesia using sufentanil to block sympathetic reactions during surgery. This decision is based on the anesthesiologist experience and not determined by the patient or procedure.
  Interventions: Procedure: opioid anesthesia
- opioid free anesthesia: anesthesia using non opioids like dexmedetomidine, lidocaine, magnesium and ketamine to block sympathetic reactions during surgery. This decision is based on the anesthesiologist experience and not determined by the patient or procedure.
  Interventions: Procedure: opioid free anesthesia

INTERVENTIONS:
Procedure: opioid anesthesia — opioid anesthesia means using sufentanil during surgery
  Groups: opioid anesthesia
Procedure: opioid free anesthesia — opioid free anesthesia means giving no opioids during surgery
  Groups: opioid free anesthesia

SUMMARY:
Opioids used intra operative increase the amount of opioids needed post operative to control post operative pain. if opioids are given post operative, we assume that more atelectasis and hypoxia takes place even after lung protective ventilation. These postoperative lower oxygen saturations will require giving more frequent oxygen therapy.

DETAILED DESCRIPTION:
This is an observational study where the attending anesthesiologist decides to use opioid free or opioid general anesthesia based on his/her expertise.

Every patient gets a lung protective ventilation and emergence from anesthesia using the principles set forward in the consensus meeting by Young C BJA 2019.

A lung recruitment followed by high PEEP is given when lung compliance decreases below 40 ML/cmH20. The lowest oxygen saturation without adding oxygen therapy is noted post extubation at moment of admission in PACU, after having given an opioid as analgesic and at moment of discharge from PACU..

If post operative satuation drops below 94% oxygen therapy is given and noted.

ELIGIBILITY:
Inclusion Criteria:

* major surgery where intubation with mechanical ventilation is required
* obese patients with BMI > 35

Exclusion Criteria:

* spontaneous breathing during procedure
* allergic to any of the drugs used in both groups
* severe liver, renal, cardiac or pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major surgery requiring intubation and mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
oxygen requirement post operative to maintain saturation above 94% | first 24 hours post operative
  oxygen saturation

SECONDARY OUTCOMES:
postoperative pain | first 24 hours post operative
  postoperative pain measured by VAS score
postoperative opioid consumption | first 24 hours post operative
  postoperative opioid consumption measured by morphine equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Marco Lanckneus, MD, Study Director — AZ Sint-Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No